CLINICAL TRIAL: NCT03281356
Title: Text Messaging Pilot Study to Encourage Shared Reading Among a Sample of Urban Parents.
Brief Title: Text Messaging Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro20170000402
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Literacy
Keywords: Pilot Study; Early childhood development
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Participants will receive a total of 8 text messages during a 4 week period.

SUMMARY:
This pilot study aims to assess the acceptability, feasibility, and preliminary effectiveness of text messages designed to encourage shared reading among urban parents. We hypothesize that parents will report reading more often to their children after receiving the text messages.

DETAILED DESCRIPTION:
This is a single arm, pilot study. The participants enrolled will receive two text messages per week for a 4 week period (a total of 8 messages). At the end of the study period we will assess change in number of reading occurrences using a validated measure. Parents will also complete a brief acceptability survey.

ELIGIBILITY:
Inclusion Criteria:

1. Preferred language either English or Spanish,
2. Parent or legal guardian,
3. Age ≥ 18,
4. Willing to accept text messages

Exclusion Criteria:

1. Individuals unable to provide consent
2. Individuals who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Acceptability Survey | Visit 2 (1 month)
  Three questions on the participants feedback on the program.

SECONDARY OUTCOMES:
Stim Q Survey | Visit 2 (1 month)
  The StimQ is a parent reported measure of the cognitive home environment

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States